CLINICAL TRIAL: NCT04024631
Title: Phenotyping Children and Adults With Possible High or Low Genetic Risk for Type 2 Diabetes
Brief Title: Phenotyping Genetic Risk for Type 2 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Jessica R.Wilson, MD, MS, Instructor in Medicine, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 831865
Record Dates: First submitted 2019-07-13; First posted 2019-07-18 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus, Type 2; Genetics
Keywords: polygenic risk for type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glucola; Absorptiometry, Photon

STUDY DESIGN:
Intervention Model Description: cross sectional
Masking Description: Data analyses (including by outcomes assessors and investigators) will be de-identified, and individuals performing laboratory analyses and DXA interpretation will be blinded to polygenic risk score for type 2 diabetes. Participants and nursing staff will not be informed of polygenic risk score at the time of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Phenotyping (Other): All participants will undergo a four-hour frequently sampled oral glucose tolerance test in which they will ingest a 75g glucose beverage (intervention) within five minutes and have samples collected at baseline and for four hours after.
  They will also undergo a whole body DXA (intervention) during the study day.
  Interventions: Other: 75g glucose beverage (Glucola, Trutol, or similar brand); Other: DXA, whole body

INTERVENTIONS:
Other: 75g glucose beverage (Glucola, Trutol, or similar brand) — Subjects will present fasting to the study day and ingest the glucose beverage during the oral glucose tolerance test.
Other: DXA, whole body — Subjects will undergo a whole body DXA scan for assessment of adiposity index and body fat distribution.

SUMMARY:
This study tests the hypothesis that non-diabetic individuals with a high genetic risk score for type 2 diabetes have impaired glucose tolerance and insulin resistance compared to those with a low genetic risk score for type 2 diabetes.

DETAILED DESCRIPTION:
The study team will recruit individuals based on genetic risk score for type 2 diabetes from the biobank populations who have agreed to be recontacted for future research. Each participant will undergo a frequently sampled four-hour oral glucose tolerance test and whole body DXA scan (dual-energy X-ray absorptiometry) in addition to baseline laboratory and history assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age 10-70 years
* Prior participant of the UPenn Biobank or Center for Applied Genomics Biobank and agreed to be recontacted for future research.
* Adults with BMI 25kg/m2 or higher, children and adolescents with BMI 85th percentile or higher

Exclusion Criteria:

* prior diagnosis of type 1, type 2, or secondary diabetes
* use of medications that would impact glucose and insulin response such as steroids, metformin or other anti-diabetic medication
* acute illness that may impact insulin and glucose dynamics
* pregnancy
* hypothalamic obesity or related genetic disorder of metabolism
* recent systemic chemotherapy use
* gastrointestinal impairment or surgery that may impact absorption
* anemia
* major organ system illness or any underlying condition requiring regular medication or treatment that could make implementation of the protocol or interpretation of the study results difficult
* inability to comply with study protocol

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-06-17 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Glucose response to an oral glucose load | samples will be collected over four hours and these results will be used to calculate area under the curve
  Glucose area under the curve after the 75g glucose beverage

SECONDARY OUTCOMES:
Visceral adiposity index | DXA scan will be obtained on the same day as the oral glucose test and will be completed in less than 30 minutes
  DXA whole body scan visceral adiposity index
HOMA-IR | calculated from baseline fasting insulin and glucose levels
  Insulin resistance estimate
Disposition index | samples will be collected over four hours after the 75g glucose beverage and these results will be used for mixed modeling
  product of insulin sensitivity and amount of insulin released; calculated using mixed modeling techniques

CONTACTS AND LOCATIONS:
Overall Officials: Jessica R Wilson, MD, MS, Principal Investigator — University of Pennsylvania; Lorraine Levitt Katz, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No